CLINICAL TRIAL: NCT05167513
Title: Monitoring Parameters Beyond Glycemic Control: Impact of Sitagliptin on Quality of Life in Type 2 Diabetes Patients
Acronym: DQOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-DM-002-20
Record Dates: First submitted 2021-11-29; First posted 2021-12-22 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Type 2 Diabetes; Metformin+Sitagliptin
Keywords: Quality of life; Type 2 Diabetes mellitus; Sitagliptin; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Uncontrolled Diabetes with Metformin or Metformin resistant (Experimental)
  Interventions: Drug: Metformin / Sitagliptin Oral Tablet

INTERVENTIONS:
Drug: Metformin / Sitagliptin Oral Tablet — Metformin and sitagliptin are oral diabetes medicines that help control blood sugar levels.
  Metformin works by decreasing glucose (sugar) production in the liver and decreasing absorption of glucose by the intestines. Sitagliptin works by regulating the levels of insulin your body produces after eating.
  Metformin and sitagliptin is a combination medicine that is used together with diet and exercise to improve blood sugar control in adults with type 2 diabetes mellitus. metformin and sitagliptin is not for treating type 1 diabetes.

SUMMARY:
Scarcity of local patients' quality of life data assessing diabetes treatment led us design a protocol to assess improvement in the quality of life of patients with Type II Diabetes mellitus. Quality of life measures are designed to enable patients' perspectives on the impact of health & healthcare interventions on their lives to be assessed & taken into account in clinical decision making & research. Its an open label experimental study where participants are assessed for quality of life impact over 6 months duration on Metformin + Sitagliptin therapy. Their safety and efficacy profiles will also be monitored

DETAILED DESCRIPTION:
Study Objective: To assess the changes in quality of life (QOL) in patients with type 2 diabetes mellitus receiving sitagliptin plus metformin therapy in routine care.

Study design: Open label, prospective, multicenter, experimental study.

Sample size: The sample size is 157. To overcome loss to follow-ups, total n=300 will be recruited where each site will enroll 30 patients.

Number of Site: There will be 10 sites.

Duration of study: 12 months (data lock point will be the completion of 6 months of follow-up from the time of last patient's enrollment date)

Study Treatment: Dose of Sitagliptin + Metformin (Treviamet® pharmaceutical brand used locally) :

For Sitagliptin + metformin: [50mg+500mg, 50mg+850mg, 50mg+1000mg] For Sitagliptin + metformin Extended Release (XR): [50mg+500mg, 50mg+1000mg].

Safety Assessment: Patient will be monitored for Hypoglycemia, Nausea, Vomiting, Diarrhea, Abdominal Discomfort, Flatulence, Asthenia, Indigestion Other adverse events and serious adverse events.

Follow up visits: After recruitment, patient is supposed to have three visits for follow-ups.

Visit 1: 4 to 6 weeks of initiation of therapy. Visit 02: At 12 weeks of initiation of therapy. Visit 03: At 24 weeks of initiation of therapy.

Study outcomes:

Primary (QoL outcomes): Diabetes Quality of Life assessment using DQOL-13 questionnaire.

Secondary (Safety and Efficacy outcomes): Frequency of adverse events and serious adverse events during the course of study follow-up. Change from baseline in HbA1c % and FBS (mg/dl) to the last-observation on treatment.

Ethical consideration: The ethical approval of study is taken from Pakistan Medical Association. The study will be conducted in compliance with the protocol, good clinical practices (GCP), the ethical principles that have their origin in the Declaration of Helsinki and the applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Type 2 Diabetes mellitus between 18 to 65 years
* HbA1C 7% - 10%
* who can give informed consent.
* Patient uncontrolled on metformin and lifestyle modification from at least 3 months or who are metformin resistant

Exclusion Criteria:

* type 1 diabetes
* ≥1 episode of Diabetic Ketoacidosis and/or hyperosmolar hyperglycemic state,
* ≥1 episode of severe hypoglycaemia,
* Pregnant or lactating women,
* Pancreatitis,
* any serious complications or hypersensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Diabetes Quality of Life assessment using DQOL-13 questionnaire | 6 months
  Satisfaction (6 questions) Impact (4 questions) Worry (3 questions)
  Scoring from 1 to 5 for worst to best quality at each question (low score means poor quality)
  Assessment at enrollment and follow ups (at 1st, 3rd and 6th months)

SECONDARY OUTCOMES:
Frequency of adverse events and serious adverse events during the course of study follow-up | 6 months
Change from baseline in HbA1c % and fasting blood sugar FBS (mg/dl) to the last-observation on treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mansoor Khan, Principal Investigator — PCDA; Asima Khan, Principal Investigator — PCDA
Locations (1):
- Primary Care Diabetes Association, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Diabetes Quality of Life (DQOL) scores, HbA1c, Fasting Blood Sugars (FBS) (masking patients' identity)

REFERENCES:
- [Derived] Khan A, Kanpurwala MA, Khan RA, Mahmudi NF, Lohano V, Ahmed S, Khan M, Uddin F, Ali SM, Saghir M, Baqar Abidi SH, Kamal J. Impact of Treviamet(R) & Treviamet XR(R) on quality of life besides glycemic control in type 2 DM patients. BMC Endocr Disord. 2023 Nov 8;23(1):244. doi: 10.1186/s12902-023-01492-2. PMID 37940936
- See also: Related Info — https://cardiab.biomedcentral.com/track/pdf/10.1186/1475-2840-12-35.pdf
- See also: Related Info — https://www.scielo.br/j/bjps/a/f36jWPRyjbQ9KwvFHNyn5mM/?lang=en